CLINICAL TRIAL: NCT05071625
Title: A Retrospectice Evaluation of the Feasibility and Usefulness of a Percutaneous Vertebroplasty Performed on Patients Treated With Posterior Fixation Suffering Non-union After a Traumatic Non-neurologic Vertebral Fracture
Brief Title: CT Guided Percutaneous Vertebroplasty for Vertebral Non-union Following Posterior Fixation
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21Imagerie02
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Vertebral Fracture; Vertebral Trauma
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: percutaneous vertebroplasty — percutaneous vertebroplasty under combined CT/fluoroscopy guidance for non-union after posterior fixation performed for a traumatic non-neurologic thoraco-lumbar vertebral fracture.

SUMMARY:
Traumatic thoracolumbar vertebral fractures are frequently treated with posterior fixation (PF) and vertebral augmentation, but sometimes vertebral augmentation is not performed, being judged too risky under fluoroscopic guidance alone. An adjuvant CT/fluoroscopy guided percutaneous vertebroplasty (PVP) could be an option.

The aim was to evaluate feasibility, safety and effectiveness of PVP in patients with vertebral non-union (VNU) following PF performed without concomitant vertebral augmentation.

All patients treated in our institution with PVP between July 2015-July 2020 were retrospectively reviewed. Patients treated with CT/fluoroscopy guided PVP under local anesthesia for symptomatic VNU following PF were selected. Three criteria were established to assess cement distribution, considering vertebral filling of: 1)fracture cleft, 2)anterior two-thirds of the vertebral body, 3)from superior to inferior endplates. Numeric pain rating scale (NPRS) assessing grade of discomfort (0=no pain; 10=worst pain) and complications were evaluated before and one month after PVP.

ELIGIBILITY:
Inclusion Criteria:

* PVP performed between July 2015-July 2020 under combined CT and fluoroscopy guidance;
* Previous PF for traumatic non-neurological thoracolumbar vertebral fracture;
* Imaging evidence of vertebral non-union;
* Pain and functional impairment persisting for more at least one month after PF;
* Informed patient consent for PVP procedure under CT and fluoroscopy guidance;
* Previous multidisciplinary case discussion between spine surgeons and interventional radiologists.

Exclusion Criteria:

* Age inferior to 18 years old
* Absence of complications due to orthopaedic hardware;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with a percutaneous vertebroplasty in our centre between 01/07/2015 and 01/07/2020 under combined CT/fluoroscopy guidance
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the procedure assessing consolidation and pain reduction 1 month after percutaneous vertebroplasty | 18 months
  Numeric Pain Rate Scale (from 0 to 10 points, where 0 no pain, 10 maximum pain)

SECONDARY OUTCOMES:
Technical success of the percutaneous vertebroplasty | 18 months
  criteria of cement filling rate of vertebral body established by the authors
Safety of the procedure | 18 months
  Complication rate during and after the procedure using CIRSE adverse event reports

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
no data sharing plan has been established